CLINICAL TRIAL: NCT01069432
Title: Protocol to Obtain Blood for Discovery of Novel Biomarkers and Potential Therapeutic Targets in Chronic Lymphocytic Leukemia
Status: Withdrawn | Type: Observational
Why Stopped: IRB delayed their review for an extensive period of time. Funding for this protocol is no longer available.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Christopher H. Lowrey, Professor of Medicine and of Pharmacology and Toxicology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D1019
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Normal Volunteers
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10cc of peripheral blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with CLL: Patients undergoing routine blood draws as part of their ongoing follow-up care for CLL at the Norris Cotton Cancer Center of DHMC.
  Interventions: Other: No Intervention
- Normal Volunteers: Normal volunteers who have no history of active or prior hematologic malignancy.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to collect a blood sample from patients with Chronic Lymphocytic Leukemia (CLL) and from volunteers without CLL.

DETAILED DESCRIPTION:
The blood sample will be used in the laboratory to perform focused studies on Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine blood draws as part of their ongoing follow-up care for CLL at the Norris Cotton Cancer Center of DHMC.
* Normal donors who have no history of active or prior hematologic malignancy.

Exclusion Criteria:

* Patients who have received cytotoxic drug, oral or intravenous steroid or targeted antibody therapy for their CLL, other hematologic malignancy or other disease process within the past 2 months are excluded. Use of intravenous immunoglobulin (IVIg) is not a reason for exclusion.
* Normal donors who have a history of steroid use, immunosuppression therapy or autoimmune disease are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Dartmouth-Hitchcock Medical Center's Norris Cotton Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
To identify the genes that are differentially expressed at the polysomal RNA and protein levels in human patient CLL cells (compared to normal donor lymphocytes) using high-throughput microarray approaches. | 2 Years

SECONDARY OUTCOMES:
To determine whether the novel candidate genes from Specific Aim 1 have potential roles in CLL. (Note: Specific Aim 2 does not involve human subjects research). | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Lowrey, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States